CLINICAL TRIAL: NCT05698719
Title: Validation of Angiography-based FFR as Compared to Pressure Wire-based FFR to Guide Revascularization of Intermediate Coronary Lesions in Non-culprit Vessels in Patients Presenting With ST-segment Elevation Myocardial Infarction
Brief Title: Validation of vFFR as Compared to FFR to Guide Revascularization of Non-culprit Lesions in STEMI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joost Daemen, Principal Investigator, Erasmus Medical Center
Other Study IDs: FAST STEMI II
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: ST Elevation Myocardial Infarction; Multivessel Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Pressure wire-based coronary physiology (FFR, RFR, dPR); Angiography-based coronary physiology (vFFR)
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Dermatopathia pigmentosa reticularis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients undergoing physiological assessment of a non-culprit lesion: vFFR, FFR, RFR, dPR, CFR and IMR

SUMMARY:
This prospective multicenter observational cohort study is designed to study the diagnostic performance of acute-setting angiography-based FFR (e.g. vFFR) for the physiological assessment of intermediate non-culprit lesions in STEMI patients, with acute-setting FFR and acute-setting NHPR (e.g. RFR) as the reference standards.

DETAILED DESCRIPTION:
The FAST STEMI II study is an investigator-initiated, multicenter, single-arm, observational cohort study aiming to include 111 patients presenting with ST-elevation myocardial infarction (STEMI). The study is designed to assess the diagnostic performance of acute-setting angiography-based fractional flow reserve (e.g. vessel fractional flow reserve (vFFR)) for the physiological assessment of intermediate non-culprit lesions, with acute-setting fractional flow reserve (FFR) and acute-setting non-hyperemic pressure ratio (NHPR) (e.g. resting full-cycle ratio (RFR)) as the reference standards.

Angiography-based FFR has the potential to guide complete revascularization in STEMI patients with multivessel disease, thereby reducing the need for invasive pressure wires and hyperemic agents. However, dedicated data regarding the diagnostic performance of acute-setting angiography-based FFR, with acute-setting FFR and NHPR as the reference standards, is currently lacking for this subset of patients.

Of note, FFR slightly underestimates the hemodynamic significance of non-culprit lesions in the acute setting due to microvascular constriction and a blunted hyperemic response, while NHPR slightly overestimates the functional lesion significance. Angiography-based fractional flow reserve is not affected by changes in the microvasculature. Potential discrepancies between acute-setting angiography-based FFR, FFR and NHPR might be explained by the microvascular state, expressed as coronary flow reserve (CFR) and the index of microvascular resistance (IMR).

Main objectives:

1. To study the diagnostic performance of acute-setting vFFR for the physiological assessment of intermediate non-culprit lesions in STEMI patients, with acute-setting FFR as the reference standard.
2. To study the diagnostic performance of acute-setting vFFR for the physiological assessment of intermediate non-culprit lesions in STEMI patients, with acute-setting RFR as the reference standards.
3. To study the impact of CFR and IMR on the potential discrepancies between acute-setting vFFR, FFR and RFR.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* At least one intermediate non-culprit lesion (50-90% diameter stenosis by visual estimation or online QCA) in a non-infarct related artery (reference vessel diameter >2.00 mm) for which invasive pressure wire-based physiological assessment is deemed feasible and indicated.

Exclusion Criteria:

* Presentation with cardiac arrest or cardiogenic shock.
* Previous coronary artery bypass graft surgery or percutaneous coronary intervention involving the non-culprit vessel.
* Ostial left main or ostial right coronary artery lesion.
* Excessive overlap, foreshortening or tortuosity precluding vFFR computation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients with multivessel disease undergoing primary percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-06-22 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of acute-setting vFFR for the physiological assessment of intermediate non-culprit lesions, with acute-setting FFR as the reference standard. | Intraprocedural (0 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value acute-setting vFFR and acute-setting FFR: ≤0.80).

SECONDARY OUTCOMES:
The diagnostic performance of acute-setting vFFR for the physiological assessment of intermediate non-culprit lesions, with acute-setting RFR as the reference standard. | Intraprocedural (0 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value acute-setting vFFR: ≤0.80; acute-setting RFR: ≤0.89).
The diagnostic performance of acute-setting RFR for the physiological assessment of intermediate non-culprit lesions, with acute-setting FFR as the reference standard. | Intraprocedural (0 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value acute-setting RFR: ≤0.89; acute-setting FFR: ≤0.80).
The diagnostic performance of acute-setting vFFR for the physiological assessment of intermediate non-culprit lesions, with offline dPR as the reference standard. | Postprocedural (max. 7 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value acute-setting vFFR: ≤0.80; offline dPR: ≤0.89).
The diagnostic performance of offline vFFR for the physiological assessment of intermediate non-culprit lesions, with acute-setting FFR and RFR as the reference standards. | Postprocedural (max. 7 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value offline vFFR: ≤0.80; acute-setting FFR: ≤0.80; acute-setting RFR: ≤0.89).
The diagnostic performance of offline vFFR for the physiological assessment of intermediate non-culprit lesions, with offline dPR as the reference standard. | Postprocedural (max. 7 days)
  Diagnostic performance: sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value (ischemic cutoff value offline vFFR: ≤0.80; offline dPR: ≤0.89).
The correlation between CFR and the potential discrepancies between acute-setting vFFR, FFR and RFR. | Intraprocedural (0 days)
  The microvascular state is expressed as coronary flow reserve (CFR).
The correlation between IMR and the potential discrepancies between acute-setting vFFR, FFR and RFR. | Intraprocedural (0 days)
  The microvascular state is expressed as the index of microvascular resistance (IMR).

CONTACTS AND LOCATIONS:
Overall Officials: Joost Daemen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Erasmus University Medical Center, Rotterdam, Netherlands
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Eijk JA, Groenland FTW, Scoccia A, Ziedses des Plantes AC, Huang J, Nuis RJ, Wilschut JM, den Dekker WK, Diletti R, Kardys I, Tomaniak M, Van Mieghem NM, Daemen J. Validation of angiography-based FFR in non-culprit vessels of patients presenting with STEMI. Clin Res Cardiol. 2025 Sep 8. doi: 10.1007/s00392-025-02729-x. Online ahead of print. PMID 40924133